CLINICAL TRIAL: NCT03770377
Title: Laryngeal Adaptation for Speech and Swallowing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB Closure
Sponsor: University of Florida (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702917 -A; R01DC016275-01A1 (NIH); OCR19032 (Other: UF ID); 5R01DC016275-02 (NIH)
Record Dates: First submitted 2018-11-29; First posted 2018-12-10 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Spinocerebellar Ataxia; Cerebral Stroke; Dysphagia; Dysarthria
Keywords: speech; swallowing; rehabilitation; stroke; deglutition; dysphagia; dysarthria; laryngeal; ataxia
MeSH Terms: conditions — Stroke; Spinocerebellar Ataxias; Deglutition Disorders; Dysarthria; Speech; Laryngeal Diseases; Ataxia

STUDY DESIGN:
Intervention Model Description: A cross-sectional study design will be used to examine laryngeal adaptation across all study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Stroke without Dysarthria (Experimental): Examine laryngeal adaptation across all study groups: (1) baseline measures of speech or swallowing , (2) a clinical examination of disease/condition severity and (3) the experimental paradigm.
  Interventions: Device: Intermittent Perturbation to Continuous Perturbation; Device: Continuous Perturbation to Intermittent Perturbation
- Stroke with Dysarthria (Experimental): Examine laryngeal adaptation across all study groups: (1) baseline measures of speech or swallowing , (2) a clinical examination of disease/condition severity and (3) the experimental paradigm.
  Interventions: Device: Intermittent Perturbation to Continuous Perturbation; Device: Continuous Perturbation to Intermittent Perturbation
- SCA6 without Dysarthria (Experimental): Examine laryngeal adaptation across all study groups: (1) baseline measures of speech or swallowing , (2) a clinical examination of disease/condition severity and (3) the experimental paradigm.
  Interventions: Device: Intermittent Perturbation to Continuous Perturbation; Device: Continuous Perturbation to Intermittent Perturbation
- SCA6 with Dysarthria (Experimental): Examine laryngeal adaptation across all study groups: (1) baseline measures of speech or swallowing , (2) a clinical examination of disease/condition severity and (3) the experimental paradigm.
  Interventions: Device: Intermittent Perturbation to Continuous Perturbation; Device: Continuous Perturbation to Intermittent Perturbation
- Age-Matched Controls (Active Comparator): Examine laryngeal adaptation across all study groups: (1) baseline measures of speech or swallowing , (2) a clinical examination of disease/condition severity and (3) the experimental paradigm.
  Interventions: Device: Intermittent Perturbation to Continuous Perturbation; Device: Continuous Perturbation to Intermittent Perturbation

INTERVENTIONS:
Device: Intermittent Perturbation to Continuous Perturbation — Manipulate the Movement Planning Period (MPP), by interrupting sensory predictions by removing e-stim during the inter-trial interval (Intermittent Perturbation), followed by a washout/de-adaptation period.
  Other Names: I to C Paradigm
Device: Continuous Perturbation to Intermittent Perturbation — Manipulate the Movement Planning Period (MPP), by keep sensory input about the perturbation constant by maintaining e-stim during the inter-trial interval.
  Other Names: C to I Paradigm

SUMMARY:
This study will test laryngeal adaptation in speech and swallowing function in healthy adults, in patients with cerebral stroke, and in patients with spinocerebellar ataxia type 6. The findings from this proposal will be the first step toward implementing rehabilitation techniques that help patients to prevent speech and swallowing errors before they occur.

ELIGIBILITY:
Patient Inclusion Criteria:

All stroke and ataxia

Ataxia

* DNA diagnosis of SCA6 and phenotype consistent with the DNA diagnosis
* No recessive, X-linked or mitochondrial

Stroke

* Bilateral or unilateral middle cerebral artery (MCA) stroke
* No structural abnormalities (i.e. nodules)
* Dysphagia involving laryngeal dysfunction

Stroke and ataxia with speech and swallowing disorders

* no structural abnormalities
* dysphagia involving laryngeal dysfunction

Patient Exclusion Criteria:

* Montreal Cognitive Assess. <24
* Moderate to severe hearing loss
* Barium allergy
* Other confounding speech disorder (i.e. stuttering)
* Chemo-radiation, surgical head and neck treatment
* Smoking Hx in the past 5 yrs or >5 years at any one time
* Twenty one years of age or older
* Breathing disorders or diseases

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Laryngeal Adaptation in Speech | Day 1
  To differentiate laryngeal adaptation during speech among cerebral stroke, SCA6, and healthy controls when vocal loudness is perturbed with expiratory loading.
Laryngeal Adaptation in Swallowing | Day 1
  To differentiate laryngeal adaptation among cerebral stroke, SCA6, and healthy controls when swallowing is perturbed with neck surface electrical stimulation to restrict laryngeal elevation.